CLINICAL TRIAL: NCT01173913
Title: Weekly Administration of (bi-)Daily Oral Docetaxel in Combination With Ritonavir
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: N10BOM
Record Dates: First submitted 2010-07-30; First posted 2010-08-02 (Estimated); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Cancer
Keywords: oral docetaxel; ModraDoc; pharmacokinetics; safety; MTD; DLT
MeSH Terms: conditions — Neoplasms | interventions — Tablets

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- ModraDoc001 10 mg capsules (Experimental): The optimal dose weekly bi-daily oral docetaxel - ModraDoc001 10 mg in combination with ritonavir will be determined with a classical dose escalation design. Approximately 24 patients will be enrolled depending on required number of dose levels before MTD is reached.
  Interventions: Drug: ModraDoc001 10mg capsules
- ModraDoc003 10mg tablets and ModraDoc004 10/50 mg (Experimental): Both new oral dosage forms, ModraDoc003 10 mg tablets and ModraDoc004 10/50 mg tablets will be investigated to see whether these new formulations have comparable pharmacokinetic characteristics, in terms of systemic exposure to docetaxel, as ModraDoc001 10 mg capsule.
  Interventions: Drug: ModraDoc003 10mg tablets and ModraDoc004 10/50 mg
- ModraDoc006 10 mg tablet (Experimental): The optimal dose weekly bi-daily oral docetaxel - ModraDoc006 10 mg in combination with ritonavir will be determined with a classical dose escalation design. Approximately 24 patients will be enrolled depending on required number of dose levels before MTD is reached.
  Interventions: Drug: ModraDoc006 10 mg tablet

INTERVENTIONS:
Drug: ModraDoc001 10mg capsules — Bi-daily administration. One cycle will last 7 days
  Arms: ModraDoc001 10 mg capsules
Drug: ModraDoc003 10mg tablets and ModraDoc004 10/50 mg — The patients will receive 40 mg docetaxel and 200 mg ritonavir once daily as different dosage forms (ModraDoc001 10 mg capsules, ModraDoc003 10 mg tablets and ModraDoc004 10/50 mg tablets). Patients continue in Week 4 with 80 mg docetaxel (as ModraDoc001 10 mg capsules) in combination with 100 mg ritonavir once daily in a weekly schedule until progressive disease or adverse events, which require dose modifications or discontinuation of therapy, are observed.
  Arms: ModraDoc003 10mg tablets and ModraDoc004 10/50 mg
Drug: ModraDoc006 10 mg tablet — Bi-daily administration. One cycle will last 7 days
  Arms: ModraDoc006 10 mg tablet

SUMMARY:
Oral administration has many advantages above intravenously administrated drugs for patients. Up to now, oral administration of docetaxel as single agent has not been feasible due to low and variable bioavailability. This low systematic exposure to docetaxel can effectively be increased after co-administration of ritonavir. The department of pharmacy of the Slotervaart Hospital and Netherlands Cancer Institute developed a solid oral dosage form for docetaxel, ModraDoc001 10 mg capsules.

Two other novel dosage forms of docetaxel with improved pharmaceutical characteristics, have been developed: ModraDoc003 10 mg tablets and ModraDoc004 10/50 mg tablets. The systemic exposure after administration of those forms is now being investigated.

DETAILED DESCRIPTION:
The bioavailability of docetaxel is limited due to metabolising cytochrome P450 (CYP) enzymes, which are abundantly present in the gastrointestinal tract.

Inhibition of CYP3A4 enzymes with ritonavir (an anti-retroviral drug) has in previously conducted proof-of-concept and phase I trials, proven to enhance the bioavailability of oral docetaxel.

Oral administration of docetaxel has been investigated in five clinical trials, all initiated by the Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital (NKI-AVL). The department of pharmacy of the Slotervaart Hospital and Netherlands Cancer Institute developed a solid oral dosage form for docetaxel, ModraDoc001 10 mg capsules. This formulation has now been investigated in more than 40 patients in a first clinical study. The preliminary results with ModraDoc001 10mg are promising and a linearity between systemic exposure to docetaxel and the applied dose of ModraDoc001 10mg capsules is seen. In an attempt to further improve and prolong the systemic exposure we will explore a twice daily dosing schedule.

Two other novel dosage forms for docetaxel, ModraDoc003 10 mg tablets and ModraDoc004 10/50 mg tablets, were developed. Both are spray-dried solid dispersions of docetaxel pressed in tablets. The distinction between both is that ritonavir is included in the co-formulation of ModraDoc004 10/50 mg tablets (10 mg docetaxel and 50 mg ritonavir). Both dosage forms will be investigated in arm B to see whether these new formulations have comparable pharmacokinetic characteristics of docetaxel to the capsule formulation.

Arm A Arm A is a dose escalation study to establish the maximum tolerated dose (MTD)of weekly bi-daily ModraDoc001 10 mg capsules. This study will be done with a classical dose escalation design. The starting dose will be 40 mg BID. This dose is based on a safety of weekly 80 mg single dose in the previously conducted study.

Arm B ModraDoc003 10 mg tablets and ModraDoc004 10/50 mg tablets will be investigated in arm B to see whether these new formulations have comparable pharmacokinetic characteristics of docetaxel to the capsule formulation od ModraDoc001 10 mg.

Another part of this study is the screening for 2 different polymorphism, C1236T (for MDR1)and CYP3A4*1B. Polymorphic variants may influence the absorption and elimination of docetaxel and ritonavir.

Arm D is a dose escalation study to establish the maximum tolerated dose (MTD)of weekly bi-daily ModraDoc006 10 mg tablets. This study will be done with a classical dose escalation design. The starting dose will be 20 mg BID. This dose is based on a safety of BID weekly ModraDoc001 mg in the previously conducted arm A.

ELIGIBILITY:
Inclusion Criteria:

1. Histological or cytological proof of cancer
2. Patients for whom no standard therapy of proven benefit exist
3. Patients who might benefit from treatment with docetaxel, e.g. advanced breast, gastric, esophagus, bladder, ovarian cancer and non-small cell lung cancer, head and neck cancers, prostate cancer and carcinoma of unknown primary site.
4. Age _ 18 years
5. Able and willing to give written informed consent
6. Able and willing to undergo blood sampling for pharmacokinetics
7. Life expectancy _ 3 months allowing adequate follow up of toxicity evaluation and anti-tumor activity
8. Minimal acceptable safety laboratory values

   * ANC of _ 1.5 x 109 /L
   * Platelet count of _ 100 x 109 /L
   * Hepatic function as defined by serum bilirubin _ 1.5 x ULN, ALAT and ASAT _ 2.5 x ULN
   * Renal function as defined by serum creatinine _ 1.5 x ULN or creatinine clearance _ 50 ml/min (by Cockcroft-Gault formula).
9. WHO performance status of _ 2
10. No radio- or chemotherapy within the last 4 weeks prior to study entry (palliative limited radiation for pain reduction is allowed)
11. Able and willing to swallow oral medication

Exclusion Criteria:

1. Patients with known alcoholism, drug addiction and/or psychotic disorders in the history that are not suitable for adequate follow up
2. Women who are pregnant or breast feeding.
3. Both men and women enrolled in this trial must agree to use a reliable contraceptive method throughout the study (adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms).
4. Concomitant use of MDR and CYP3A modulating drugs such as Ca+-entry blockers (verapamil, dihydropyridines), cyclosporine, quinidine, quinine, tamoxifen, megestrol and grapefruit juice, concomitant use of HIV medications; other protease inhibitors,(non) nucleoside analoga, St. Johns wort or macrolide antibiotics as erythromycin and clarithromycin.
5. Uncontrolled infectious disease or known HIV-1 or HIV-2 type patients
6. Unresolved (>grade 1) toxicities of previous chemotherapy
7. Bowel obstructions or motility disorders that may influence the absorption of drugs
8. Chronic use of H2-receptor antagonists or proton pump inhibitors
9. Neurologic disease that may render a patient at increased risk for peripheral or central neurotoxicity
10. Pre-existing neuropathy greater than CTC grade 1
11. Symptomatic cerebral or leptomeningeal metastases
12. Evidence of any other disease, neurological or metabolic dysfunction, physical examination finding or laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or puts the patient at high risk for treatment-related complications.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2010-09 (Actual); Primary Completion 2016-10-04 (Actual); Study Completion 2017-01-26 (Actual)

PRIMARY OUTCOMES:
Number and percentage of Participants with Adverse Events | AE will be collected during the study treatment and 30 days after discontinuation of the study treatment due to disease progression or unacceptable treatment related toxicity
  The maximal tolerated dose (defined as the highest dose resulting in no more that 1/6 probability of causing a dose limiting toxicities defined in the protocol) of bi-daily ModraDoc001 10mg capsules with ritonavir will be assessed in Arm A. Weekly safety assessments for Arm A and Arm B: signs and symptoms/adverse events, physical examination, clinical laboratory tests (hematology, clinical chemistry and urinalysis), 12-lead ECG monitoring (Day 0, End of Th). The incidence of serious AEs (SAEs) and AE related to oral docetaxel and/or to ritonavir will be determined.

SECONDARY OUTCOMES:
Pharmacokinetics assessments | Day 1 of week: 1, 2 and 3
  The PK of bi-daily ModraDoc001 10mg, ModraDoc003 10mg tablets both in combination with ritonavir capsules and ModraDoc004 10/50mg tablets will be determed using non-compartmental methods and compartmental methods using NONMEM. Correlation between PK data and toxicity are subsequently analyzed for their significance.
Number and percentage of Participants with Adverse Events | during the study treatment and 30 days after the study discontinuation
  Weekly safety assessments for Arm B (administration of ModraDoc003 10mg capsules and ritonavir and ModraDoc004 10/50 mg tablets) are: signs and symptoms/adverse events, physical examination, clinical laboratory tests (hematology, clinical chemistry and urinalysis), 12-lead ECG monitoring (Day 0, End of Th). The incidence of serious AEs (SAEs) and AE related to oral docetaxel and/or to ritonavir will be determined.
Radiological antitumor activity | at least every six weeks
  Tumor measurement according to RECIST
Pharmacogenetic sampling | Day 1 - predose
  To establish the effect of functional genetic polymorphisms, C1236T (for MDR1) and CYP3A4*1B, on pharmacokinetics of orally administered docetaxel.

CONTACTS AND LOCATIONS:
Overall Officials: JHM Schellens, MD, PhD, Principal Investigator — The Netherlands Cancer Institute
Locations (1):
- Netherlands Cancer Institute - Antoni van Leeuwenhoek Hospital, Amsterdam, Netherlands

REFERENCES:
- [Derived] Vermunt MAC, van der Heijden LT, Hendrikx JJMA, Schinkel AH, de Weger VA, van der Putten E, van Triest B, Bergman AM, Beijnen JH. Pharmacokinetics of docetaxel and ritonavir after oral administration of ModraDoc006/r in patients with prostate cancer versus patients with other advanced solid tumours. Cancer Chemother Pharmacol. 2021 Jun;87(6):855-869. doi: 10.1007/s00280-021-04259-5. Epub 2021 Mar 20. PMID 33744986
- See also: Article on the study — https://www.ncbi.nlm.nih.gov/pubmed/29031170